CLINICAL TRIAL: NCT02988037
Title: Adapted Dialectical Behaviour Therapy for Adolescents With Deliberate Self-Harm: A Pre-post Observational Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Darren Courtney, Assistant Professor in the Department of Psychiatry, University of Ottawa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G6302346
Record Dates: First submitted 2016-11-27; First posted 2016-12-09 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Deliberate Self Harm; Borderline Personality Disorder
MeSH Terms: conditions — Self-Injurious Behavior; Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A-DBT-A (Experimental): Began Adapted Dialectical Behaviour Therapy for Adolescents
  Interventions: Behavioral: A-DBT-A

INTERVENTIONS:
Behavioral: A-DBT-A — Adapted Dialectical Behaviour Therapy for Adolescents

SUMMARY:
The investigators conducted a pre-post naturalistic study regarding changes observed associated with a 15-week course of an adapted form of dialectical behaviour therapy for adolescents. We measured frequency of self-harm prior to treatment and after treatment using the Self-Injurious Thoughts and Behaviors Interview. We also measured changes using the Suicide Ideation Questionnaire, Life Problems Inventory, Resiliency Scale for Children and Adolescents.

ELIGIBILITY:
Inclusion Criteria:

* features of Borderline Personality Disorder (BPD) and recent history of self-injurious thoughts or behaviours.

  1. meeting criteria for BPD or for subsyndromal variants of BPD, and (2) self-injurious thoughts and behaviours defined as: (a) a score > 30 on the Suicidal Ideation Questionnaire (SIQ) OR (b) Deliberate Self-harm in the 4 months prior to treatment

Exclusion Criteria:

* severe substance use (where residential treatment would be indicated), florid psychosis and developmental delay

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2012-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Deliberate Self-harm | 15 weeks
  Self-Injurious Thoughts and Behaviors Interview was performed by clinicians. Using the scale the investigators rated the frequency of deliberate self-harm of participants (with or without suicidal intent) as "most days", "twice or more per week", "once or more per week", "less than once per week", "less than once per 2 weeks" and "less than once a month" or "no self-harm" in the 4 month interval prior to treatment and the 4 month interval during treatment.

SECONDARY OUTCOMES:
Suicidal Ideation Questionnaire | 15 weeks
  Self-report measure was requested a baseline and end of treatment to measure the severity of suicidal ideas.
Life Problems Inventory | 15 weeks
  Symptoms of Borderline Personality Disorder were measured by a self-report form at baseline and post-treatment.
Resiliency Scales for Children and Adolescents | 15 weeks
  RSCA is a self-report measure that was performed at baseline and post-treatment.
Attrition from therapy | 15 weeks
  If participants missed 4 or more individual therapy sessions; OR 4 or more group sessions, they were considered to have "dropped out" of therapy.

IPD SHARING:
Plan to Share IPD: No